CLINICAL TRIAL: NCT05133141
Title: A Prospective, Single-Arm, Multi-Center Study of the ECHELON ContourTM Curved Cutter Stapler Device in Colorectal Procedures
Brief Title: A Study of the ECHELON Contour Curved Cutter Stapler Device in Colorectal Procedures
Status: Terminated | Type: Observational
Why Stopped: This clinical study was terminated due to low recruitment.
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC202102; ESC202102 (Other: Ethicon Endo-Surgery)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Echelon Contour: This prospective study will include the participants who plan to have an elective colorectal surgical procedure and collect clinical data in a post-market setting. Investigators will perform each procedure using the device in compliance with their standard surgical approach and the Echelon Contour instruction for use (IFU).
  Interventions: Device: Echelon Contour

INTERVENTIONS:
Device: Echelon Contour — There is no intervention, beyond necessary clinical care, in this study. Echelon Contour is used for transection and resection in colorectal surgical procedures per its instructions for use (IFU).

SUMMARY:
The purpose of this study is to prospectively generate device-specific clinical data related to the performance of Echelon Contour per its instructions for use (IFU).

ELIGIBILITY:
Inclusion Criteria:

* Elective colorectal procedure where Echelon Contour is planned to be used for transection and resection of the colon
* Willingness to give consent and comply with all study-related evaluations and visit schedule. If the participant is less than (<) 18 years of age, the participant's parent/legal guardian must be willing to give permission for the participant to participate in the study and provide written Informed Consent for the participant. In addition, assent must be obtained from pediatric participants who possess the intellectual and emotional ability to comprehend the concepts involved in the study. If the pediatric participant is not able to provide assent (due to age, maturity and/or inability to intellectually and/or emotionally comprehend the study); the parent/legal guardian's written Informed Consent for the participant will be acceptable for the participant to be included in the study
* Anatomical region must be of sufficient size for the device to be used

Exclusion Criteria:

Preoperative

* Females who are pregnant
* Physical or psychological condition which would impair study participation
* Participant previously enrolled into the study (example: participant enrolled for Hartmann's procedure then cannot be reenrolled for the Hartmann's reversal)

Intraoperative

- Study device use not attempted

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who plan to have an elective colorectal surgical procedure will be included.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Echelon Contour Success | interoperative
  Echelon Contour success based on surgeon responses on question 1 in the surgeon reported outcome measures (SROM) will be reported. Surgeon will be asked to choose option "Yes" or "No" for following question: Did Echelon Contour provide acceptable performance considering other therapeutic alternatives?

SECONDARY OUTCOMES:
Number of Participants with Device-related Adverse Events (AEs) | 28 days post-procedure
  An AE is defined as any untoward medical occurrence, regardless of its relationship to the study device or the study procedure. An untoward medical occurrence includes any new, undesirable medical experience or worsening of a pre-existing condition, which occurs throughout the duration of the clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon Endo-Surgery Clinical Trial, Study Director — Ethicon Endo-Surgery
Locations (2):
- United States (2):
  - Baylor Scott and White, St Louis, Missouri
  - Washington University, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Rai P, Johnston SS, Chaudhuri R, Naoumtchik E, Pollack E. Association of Complications with Healthcare Utilization and Hospital-Borne Costs Among Patients Undergoing Open Low Anterior Resection Using Curved Cutter Staplers. Med Devices (Auckl). 2021 Mar 31;14:87-95. doi: 10.2147/MDER.S298975. eCollection 2021. PMID 33833593
- [Background] Giustina A, Bevan JS, Bronstein MD, Casanueva FF, Chanson P, Petersenn S, Thanh XM, Sert C, Houchard A, Guillemin I, Melmed S; SAGIT Investigator Group. SAGIT(R): clinician-reported outcome instrument for managing acromegaly in clinical practice--development and results from a pilot study. Pituitary. 2016 Feb;19(1):39-49. doi: 10.1007/s11102-015-0681-2. PMID 26377024